CLINICAL TRIAL: NCT01859845
Title: Melanoma Simulation Model With Smartphone Devices: Training Physicians to Perform Opportunistic Surveillance for Early Detection of Melanoma
Brief Title: Melanoma Simulation Model With Smartphone Devices: Training Physicians for Early Detection of Melanoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, June Robinson, Research Professor of Dermatology, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: STU00077615
Record Dates: First submitted 2013-05-20; First posted 2013-05-22 (Estimated); Last update posted 2014-08-01 (Estimated); Status verified 2014-07

CONDITIONS: Melanoma
Keywords: Melanoma; Opportunistic surveillance; Melanoma simulation model; Smartphone devices
MeSH Terms: conditions — Melanoma | interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Study Arm (No Intervention): The control participants will first interact with the simulated melanoma back model to learn clinical unaided visual inspection skills and then view a passive image projected onto a screen for dermoscopy learning. Remediation of inappropriate clinical decisions will be carried out by the research coordinator and is based on predefined feedback consistent across both arms of the study. Along with the projected images, the coordinator will provide each control participant with worksheets for the clinical Asymmetry, Border, Color, Diameter (ABCD) and Dermoscopy 3-point check list. A copy of the completed worksheet will be made at the end of the workshop.
- smartphone (Experimental): Each participant in the educational intervention arm will have access to a smartphone with a preloaded android software package. The smartphone software allows the participant to visualize a dermoscopic image of the pigmented lesion at the surface of the simulated melanoma model. Participants are given the freedom to navigate through the program via the smartphone to learn at their own pace with reinforcement of correct clinical management decisions and correction of weaknesses. The software content is limited to the dermoscopy information available to the positive control arm through the coordinator and the dermoscopic images projected onto the screen, thus a comparison of retention rates across both arms is possible.
  Interventions: Other: Smartphone

INTERVENTIONS:
Other: Smartphone — Our team of dermatologists and biomechanical engineers led by the PI developed a simulation skills training prototype device using a smartphone. Software was developed to teach dermoscopic evaluation of pigmented lesions using the "three-poin checklist of dermoscopy". The software used in the smartphone presentation of the educational intervention also provides a decision tree of clinical management options and best-practices feedback. No patients are involved in this research.
  Other Names: educational intervention
  Arms: smartphone

SUMMARY:
The specific aim of this study is to determine if interactive touchscreen-based learning with deliberate practice modules can enhance the retention of life-saving medical skills when incorporated into medical training curricula. We will analyze the retention and confidence of screening skills by comparing outcomes on pretest and posttest in each arm.

DETAILED DESCRIPTION:
Age-adjusted melanoma incidence among Caucasians has risen from 7.5 to 21.9 cases per 100,000 representing an increase of nearly 200% over 30 years. In contrast to other cancers (i.e. colorectal, prostate, cervical), melanoma is detected by intentional visual skin inspection. Intentional screening is the deliberate visual inspection of all cutaneous surfaces. However, fewer than 30% of primary care physicians (PCPs) reported training in skin cancer during their medical education. Early detection of melanoma by PCPs cannot be expected to improve without addressing both the PCPs' lack of training and their low confidence in examination skills pertaining to pigmented lesion exams. A focused intervention is required to improve PCPs' early detection of melanoma and mitigate the near-term consequences of an aging US population.

Opportunistic surveillance requires skills in both unaided visual inspection of the skin and in dermoscopy of lesions. Dermoscopy-a hand-held magnifying device that assists with diagnosis-reduces the number of unnecessary biopsies and improves the clinical sensitivity of diagnosing melanoma. Studies show that Australian PCPs trained to use a "three-point checklist of dermoscopy," developed biopsy ratios of benign to malignant lesions of 8:1 in the general population, which is comparable to dermatologists using dermoscopy. In 2009, the American Academy of Family Physicians held their first dermoscopy course at their Annual Scientific Meeting, and there is continuing demand for similar courses. By making dermoscopy customary for PCPs, PCPs will be able to detect melanomas opportunistically and render care to the at-risk population of elderly for whom they provide care. Smart-touchscreen technologies can potentially provide a safe environment for medical trainees to learn procedural and screening skills that are rarely available opportunities in the clinic. As such, these technologies may lead to better health outcomes in future populations.

In this study, eighty 3rd year medical and thirty 1st year physician's assistant students participate in a visual screening and dermoscopy curriculum aimed at improving the retention rate of the learned clinical skills. After a didactic lecture on melanoma screening, participants are randomized to either a control or an experimental study arm for the clinical skills workshop. The control arm represents our previously published clinical skills training workshop (IRB STU 0002705) in which participants interact with a simulated patient model presenting with pigment lesions and review dermoscopy images on a projector screen. In the experimental arm, the projector-based learning approach is replaced with a handheld touchscreen device (smartphone) preloaded with interactive melanoma screening tutorial. The smartphone provides instant feedback and remediation of improper clinical management decisions. Across both groups, all learning content remains similar. Further deliberate practice questions provided to the control arm are standardized while the experimental arm's questions are individualized based on weaknesses determined in the smartphone software.

ELIGIBILITY:
Inclusion Criteria for Evaluation of the smartphone-based dermoscopy prototype device:

* Thirty 4th year medical students and 2nd year physician assistant (PA) students with previous experience with the Melanoma Simulation Model of the back (IRB STU00025072)

Inclusion Criteria for teaching and testing sessions with medical students and physician assistant students:

* Eighty third-year medical students and thirty PA students

Exclusion Criteria:

* Those not meeting the above inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2013-04; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Evaluation of medical student's abilities to select pigmented lesions for review with dermoscopy on pre-didactic lecture test, pre-skills workshop test, and post-educational intervention test | Two weeks post initial didactic education
  Retention will be measured using the percent of correctly identified benign nevi, clinically suspicious lesions, and melanomas identified by unaided visual inspection and the percent of correctly identified "benign" or "refer" lesions on dermoscopy images. The biopsy ratio of benign to malignant lesions will be also be assessed to determine the sensitivity and specificity outcomes of both study arms. Other outcomes measured are the confidence with identifying melanoma, attitudes toward melanoma screening, and recall of screening rules by participants. The rates of retention in both study arms will be compared on pre-workshop test and the post-test to determine if simulation learning modules positively impact learning and retention of skin screening.

CONTACTS AND LOCATIONS:
Overall Officials: June K Robinson, MD, Principal Investigator — Northwestern University Department of Dermatology
Locations (1):
- Northwestern University Department of Dermatology, Chicago, Illinois, United States